CLINICAL TRIAL: NCT05106491
Title: Evaluating the Efficacy and Safety of the Synchronized Cardiac Support Treatment with the Icor Kit in Patients with Cardiogenic Shock - a Pivotal Study (Pulse SE)
Brief Title: Efficacy and Safety of Synchronized Cardiac Support in Cardiogenic Shock Patients
Acronym: PulseSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xenios AG (Industry)
Responsible Party: Sponsor
Organization: Fresenius Medical Care Deutschland GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CS-SCS-01-DE
Record Dates: First submitted 2021-10-05; First posted 2021-11-03 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation; ECLS; VA ECMO
Keywords: Cardiogenic Shock; Extracorporeal Membrane Oxygenation; Synchronized Cardiac Support; ECLS; VA ECMO
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- venoarterial extracorporeal membrane oxygenation (VA ECMO) for cardiocirculatory stabilization (Other): Patients with cardiogenic shock, requiring a venoarterial extracorporeal membrane oxygenation (VA ECMO) for cardiocirculatory stabilization will be treated with Synchronized Cardiac Support (SCS).
  Interventions: Device: Synchronized Cardiac Support with the icor kit

INTERVENTIONS:
Device: Synchronized Cardiac Support with the icor kit — Patients with cardiogenic shock, requiring a venoarterial extracorporeal membrane oxygenation (VA ECMO) for cardiocirculatory stabilization will be treated with Synchronized Cardiac Support (SCS).
  Other Names: Synchronized Cardiac Support (icor)

SUMMARY:
The study aims to investigate the safety and efficacy of the Synchronized Cardiac Support treatment wit the icor kit and the Xenios console with modified sensor box ECG and Software Version 3.2.4

DETAILED DESCRIPTION:
The current study hypothesizes that The SCS treatment with the icor kit provides sufficient support for cardiocirculatory function as indicated by a significant lactate reduction 24 hours on SCS treatment versus before treatment start.

Patients with cardiogenic shock, requiring a venoarterial extracorporeal membrane oxygenation (VA ECMO) for cardiocirculatory stabilization will be treated with Synchronized Cardiac Support.

Synchronized Cardiac Support describes an electrocardiogram (ECG)- triggered pulsatile VA-ECMO based on R-wave detection. During diastole the pump speed and thus the flow is increased and during systole the pump flow is been set on a relative minimum. This provides a mechanical circulatory support pulse with oxygenated blood during diastole.

The Synchronized Cardiac Support Treatment is used in a standard VA ECMO configuration by two femoral single vessel cannulas. Patients following cardiac resuscitation will undergo targeted temperature management 32- 36°C according to guideline.

The Duration of Treatment can be up to 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed and dated by study patient/legal representative and investigator/authorised physician
2. Minimum age of 18 years
3. Patients in cardiogenic shock
4. Cardiogenic shock is defined as:

   1. Systolic blood pressure < 90 mmHg for at least 30 min
   2. Inotropes and/or vasopressors are needed to maintain systolic blood pressure > 90 mmHg
   3. Clinical signs of heart insufficiency with pulmonary congestion
5. Signs of end organ hypoperfusion with at least one of the following criteria:

   1. Cold, damp skin or extremities
   2. Oliguria (≤ 30 mL/h)
6. Serum lactate > 3.0 mmol/L

Exclusion Criteria:

1. In case of female patients: pregnancy or lactation period
2. Participation in an interventional clinical study during the preceding 30 days
3. Previous participation in the same study
4. Age > 85 years
5. Cardiac arrest out of hospital with return of spontaneous circulation (ROSC) > 30 min
6. No flow time > 5 min
7. Mechanical causes for cardiogenic shock (ventricular septal defect of papillary muscle rupture)
8. Non-cardiogenic causes of shock (bradycardia, sepsis, hypovolemia, etc.)
9. Fever (Body temperature > 38.0 °C) or other evidence of sepsis
10. Onset of cardiogenic shock > 6 h before enrolment
11. Lactate > 16 mmol/L
12. Severe peripheral arterial occlusive disease precluding insertion of femoral arterial or venous catheters
13. Contra-indications for anticoagulation
14. Contra-indication for VA ECMO, e.g. unrecoverable heart and not a candidate for transplant or VAD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Cardiocirculatory stabilization and end-organ perfusion | up to 14 days
  measured by the Change in Lactate Level

SECONDARY OUTCOMES:
Cardiocirculatory stabilization and end-organ perfusion | up to 14 days
  measured by the following parameter: Mean Arterial Pressure, Catecholamine Support, Cardiac Index, Cardiac Output and Cardiac Afterload
Maintain gas exchange | up to 14 days
  measured by the following parameter: Blood Gas Analysis and Mechanical Ventilation
Extracorporeal Life Support (ECLS) Performance | up to 14 days
  measured by the following parameter: Blood Flow, Blood Pressure, Synchronization of the patient's heartbeat, Intra-hospital transportation
Maintain renal function | up to 14 days
  measured by the following parameter: Fluid Balance, Renal Replacement Therapy, Creatinine and eGRF
Thermoregulation | up to 14 days
  measured by the the Body Temperature

OTHER OUTCOMES:
Safety Variables | up to 14 days
  1. Severe adverse events, i.e. Hemolysis Bleeding
  2. Severe adverse device events

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Voigt, Dr., Principal Investigator — Elisabeth-Krankenhaus Essen
Locations (2):
- Germany (2):
  - Krankenhaus Buchholz und Winsen gGmbH, Buchholz
  - Elisabeth-Krankenhaus Essen GmbH, Essen